CLINICAL TRIAL: NCT06681376
Title: Enhancing the Emergency Department Experience for Older Adults: Study Protocol for the Implementation of a Comfort Menu and Cart
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Pedro Kallas Curiati, Principal Investigator, Hospital Sirio-Libanes
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AVAP-NG 3776
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Emergency Department Patient; Comfort
Keywords: comfort cart; patient experience; older adult; emergency department
MeSH Terms: conditions — Emergencies | interventions — Cocaine- and Amphetamine-Regulated Transcript Protein

STUDY DESIGN:
Intervention Model Description: This study will utilize a quasi-experimental, before-and-after design.
Who Masked: Outcomes Assessor
Masking Description: A research assistant, blinded to the initial assessment and ED care details, will conduct a phone interview 30 days (± 2 days) post-initial assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-intervention (No Intervention): Usual ED care
- Post-intervention (Experimental): Comfort menu and cart implemented
  Interventions: Other: Comfort menu and cart

INTERVENTIONS:
Other: Comfort menu and cart — The comfort menu and cart will be implemented after the pre-intervention data collection phase is completed. The menu will list the items available on the cart and will be presented to eligible patients in printed or digital format (on a tablet). The cart will be placed in an easily accessible area within the ED. Approximated retail prices have been previously reported.
  Comfort Cart Contents:
  * Hot and cold packs;
  * Extra blanket and pillow;
  * Face towel;
  * Gloves and hat;
  * Personal hygiene kit;
  * Items for distraction;
  * Items to enhance communication.
  Comfort Menu Options:
  * Physiotherapy assessment;
  * Conversation with chaplain, concierge, or social worker;
  * List of resources for older adults needing community services;
  * Home care assistance.
  Arms: Post-intervention

SUMMARY:
Introduction: The aging of the population is a global phenomenon, with projections indicating a significant increase in the proportion of individuals aged 65 years and older by 2050. This demographic shift requires adapting emergency department (ED) services to meet the specific demands of older patients, who often present with multiple comorbidities and face challenges such as sensory and cognitive difficulties. EDs, traditionally designed for acute illness and injury management, may not be adequately equipped to meet the unique needs of this vulnerable population. This can result in suboptimal patient experiences, prolonged ED stays, increased hospitalizations, and poorer outcomes.

Methods: This study protocol outlines a before-and-after study to evaluate the impact of implementing a comfort menu and cart on the experience and outcomes of older patients treated in the ED. The study will be conducted in the ED of Hospital Sírio-Libanês (HSL), a tertiary private hospital in São Paulo, Brazil. Patients aged 65 and older who presented to the ED will be eligible for inclusion. Participants will be recruited in two phases: pre-intervention and post-implementation of the comfort menu and cart. Data will be collected through patient and staff interviews, chart reviews, and a 30-day follow-up interview. Patient experience, staff experience, length of hospital stays, hospital costs, ED readmissions, falls, delirium incidence, quality of life, functional status, cognitive performance, and mortality will be assessed.

Ethics and dissemination: Ethical approval for this study has been granted by the Institutional Review Board of HSL. All participants, or their legal representatives for those with cognitive impairment, will provide written informed consent before any study procedures are initiated. The consent process has been designed keeping the study hypothesis blind by not revealing the outcomes that will be measured after the comfort cart intervention. The results will be shared with the academic community through peer-reviewed publications and presentations at relevant conferences to inform future clinical practice and research.

Expected Results: A positive impact of implementing the comfort menu and cart in the ED is expected on patient-centered outcomes. Improvements in the experience of older patients and medical and multidisciplinary staff are anticipated, and improvements in other exploratory outcomes, such as length of hospital stay, hospital costs, readmissions, falls, delirium incidence, quality of life, functionality, and cognitive performance, will be explored.

ELIGIBILITY:
Inclusion Criteria:

* ED attendance at Hospital Sírio-Libanês (HSL), São Paulo, Brazil.
* Age ≥ 65 years.
* Capacity to consent and respond to the interview or the presence of a companion capable of doing so.

Exclusion Criteria:

* Decline to participate in the study or use the comfort menu and cart.
* Absence of a companion able to consent to study participation and provide necessary information for patients with altered mental status or cognitive impairment.
* Decreased level of consciousness.
* Hemodynamic instability.
* Acute respiratory failure.
* Inability to be contacted by phone for the follow-up interview.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Experience of older patients treated in the ED | Baseline assessment during ED stay
  Likert scale and brief questionnaire adapted from previous studies

SECONDARY OUTCOMES:
Experience of medical and multidisciplinary staff involved in caring for older patients treated in the ED | 3 months pre- and post-intervention, concurrent with patient inclusion
  The interview will follow the standardization of the original comfort cart validation study, using a Likert scale.

OTHER OUTCOMES:
Length of hospital stay | From the index ED admission to hospital discharge
  Duration of the patient stay from ED admission to hospital discharge
Hospital costs | From the index ED admission to hospital discharge
  All costs associated to patient care during the index ED visit and hospital stay
Readmissions | 30 days
  Rate of ED and hospital readmissions after de index ED visit
Falls | 30 days
  Rate of falls after hospital discharge
Delirium incidence | 30 days
  Assessed using the Family Confusion Assessment Method (FAM-CAM)
Quality of life | 30 days
  Assessed using the Euro Quality of Life Instrument - 5D. t encompasses five health domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is classified into three levels: no problems (1 point), some problems (2 points), and extreme problems (3 points). Additionally, it includes a self-assessment of health on a visual analog scale (VAS), ranging from 0 (worst possible health) to 100 (best possible health), resulting in 243 out of 3125 distinct health states.
Functionality - Basic activities of daily living | 30 days
  Assessed using the Katz Index and Barthel Indexes. The Katz Index assesses self-care in Activities of Daily Living, with a score ranging from 0 (total independence) to 6 (total dependence). The Barthel Index measures functional independence in personal care and mobility, with a score from 0 to 100, classifying dependence from total to minimal.
Functionality - Instrumental activities of daily living | 30 days
  The Lawton and Brody scale assesses seven Instrumental Activities of Daily Living, with scores ranging from 9 to 27, classifying dependence from total to mild.
Cognitive performance | 30 days
  Assessed using the 10-Point Cognitive Screener. With a score ranging from 0 to 10, it classifies cognitive performance as normal (≥8), possible cognitive impairment (6-7), or probable cognitive impairment (0-5), with adjustments for education level.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro K Curiati, M.D., Ph.D., Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Patient confidentiality

REFERENCES:
- [Derived] Ferreira SA, Bellolio F, Bower SM, Penna LF, Marion MAL, Aliberti MR, Avelino-Silva TJ, Morinaga CV, Curiati PK. Enhancing the emergency department experience for older adults: Study protocol for the implementation of a comfort menu and cart. PLoS One. 2025 Dec 4;20(12):e0332773. doi: 10.1371/journal.pone.0332773. eCollection 2025. PMID 41343524